CLINICAL TRIAL: NCT03002363
Title: The Effects of Video Modeling of Audiological Testing on Pediatric Patient Compliance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Megan Roberts, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00203250
Record Dates: First submitted 2016-12-09; First posted 2016-12-23 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Autism
Keywords: autism; audiology; video modeling; testing compliance
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video Modeling Intervention (Experimental): The intervention group receives a video that is a behavior modeling video that walks through the entire audiological evaluation. It also includes tips for caregivers to practice with their child before the appointment.
  Interventions: Behavioral: Video Modeling Intervention
- Placebo Video (Placebo Comparator): The other video is a placebo video that discusses hearing, listening and ears, that does not discuss tips for caregivers to practice with their child before the appointment. The placebo video is not related to the audiological evaluation.
  Interventions: Behavioral: Placebo Video

INTERVENTIONS:
Behavioral: Video Modeling Intervention — Prior to arrival of the audiological evaluation, the child and caregiver will be required to watch one of two videos created by the research personnel. One video, the intervention video, is a behavior modeling video walking through the entire audiological evaluation. It also includes tips for caregivers to practice with their child before the appointment. The other video is a placebo video that discusses hearing, listening and ears, that does not discuss tips for caregivers to practice with their child before the appointment. The placebo video is not related to the audiological evaluation.
  Arms: Video Modeling Intervention
Behavioral: Placebo Video — The other video is a placebo video that discusses hearing, listening and ears, that does not discuss tips for caregivers to practice with their child before the appointment. The placebo video is not related to the audiological evaluation.
  Arms: Placebo Video

SUMMARY:
The purpose of the current study is to determine if pre-exposure through video modeling will enhance testing compliance in a population of children who are receiving a diagnostic evaluation for Autism.

DETAILED DESCRIPTION:
The purpose of the current study is to determine if pre-exposure through video modeling will enhance testing compliance in a population of children who are receiving a diagnostic evaluation for Autism. Another purpose of this study is to determine if pre-exposure to the test setting can increase the compliance on individual test measures. To test the central hypothesis and accomplish the study objective, 2 aims guide the proposed study.

1. Determine the extent to which pre-exposure to expectations and tasks that occur during the audiological evaluation will increase audiological testing compliance. Hypothesis: Children receiving the intervention video, which will model what they will experience during the audiological evaluation, will show greater compliance during the evaluation than children who receive the placebo video.
2. Determine the extent to which enhanced testing compliance will increase the number of test measures obtained during an audiological evaluation. Hypothesis: Children who are more compliant during the audiological evaluation will allow the audiologist to obtain more test measures in a single appointment than the children who are less compliant.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Child must have chronological age of less than 36 months
* Participation in the Northwestern University Center for Audiology, Speech, Language, and Learning (NUCASLL) Developmental Diagnostic Program (DDP)
* A parent or caregiver who is willing to watch the intervention video, bring the child to/ participate in the audiological evaluation, and fill out a brief survey prior to and following the appointment, and
* Parent must understand English and speak English to their child.

Exclusion Criteria:

* None

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Compliance to audiology tests (% of audiology tests completed during an audiology session) | Immediately following appointment (same day as appointment)
  Compliance to the following audiology test battery: Otoscopy, Speech Awareness Threshold, Pure Tone Testing, Distortion, Product Otacoustic Emissions, Tympanometry. Compliance is measured as either "yes" or "no" to each of the tests in order to measure how many audiology tests are completed at the visit. The individual test units do not matter for the overall compliance of the visit.

SECONDARY OUTCOMES:
Parent stress | Immediately before and immediately after audiology appointment (same day as appointment)
  PI developed form regarding parent perception

CONTACTS AND LOCATIONS:
Overall Officials: Megan Y Roberts, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Clinic for Audiology, Speech, Language, and Learning, Evanston, Illinois, United States